CLINICAL TRIAL: NCT06251323
Title: Implementing Scalable, PAtient-centered, Team-based, Technology-enabled Care for Adults With Type 2 Diabetes (iPATH)
Acronym: iPATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Ohio State University (Other); Harvard School of Public Health (HSPH) (Other); Impactivo, LLC. (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sara Singer, Professor of Health Policy, of Medicine (Primary Care & Population Health), by courtesy, of Organizational Behavior at the Graduate School Of Business and Senior Fellow, by courtesy, at The Freeman Spogli Institute For International Studies, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 72410; 1R01MD017870-01A1 (NIH)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wave 1 Clinics (Experimental): Clinics will have data evaluated for up to 3 years. Wave 1 clinics will begin the iPATH practice transformation in Year 1.
  Interventions: Other: iPATH implementation approach
- Wave 2 Clinics (Experimental): Clinics will have data evaluated for up to 3 years. Wave 2 clinics will begin the iPATH practice transformation in Year 2.
  Interventions: Other: iPATH implementation approach

INTERVENTIONS:
Other: iPATH implementation approach — A multi-level, multi-component, customized, standardized, technology enabled, person-centered, and team-based care practice transformation strategy.

SUMMARY:
Sixteen institutions will be selected from a HRSA uniform data system and have data collected for up to 3 years. Eight institutions will begin the iPATH practice transformation during year one, the other eight institutions will begin iPATH in year two. FQHC administrators, clinicians and staff will be enrolled to participate in the iPATH transformation in their clinic and will participate in qualitative interviews. Patient HbA1c data from the clinics will be collected for comparative data analysis during each year of the study.

DETAILED DESCRIPTION:
A collaborative network of research teams from Stanford, Harvard, The Ohio State University, and Impactivo, LLC propose practice-relevant research focused on diabetes care in federally qualified health centers (FQHCs). Some 37.3 million Americans have type 2 diabetes. FQHCs are an important source of diabetes care for one in ten Americans and shoulder a higher prevalence of diabetes (21% FQHC, 11% U.S.), offering a promising venue for innovating in diabetes care. The iPATH project will refine and implement an approach to practice transformation originally conceived to support FQHCs' pursuit of National Committee for Quality Assurance recognition as patient-centered medical homes. A pilot demonstrated significant decreases (average 31% reduction) in poorly controlled diabetes (A1c>9%) among patients at 7 clinics affiliated with an FQHC in Puerto Rico in 2017-20. Improvements in patients' diabetes control were sustained pre- to post- Covid-19 pandemic.

Aim 1. Refine the iPATH implementation approach by identifying organizational conditions and processes at FQHCs that promoted or impeded the effectiveness of type 2 diabetes care. Research teams will simultaneously conduct 12 in-depth regional case studies, enabling contrast between FQHCs considered high-performing and low-performing for diabetes control. Teams will identify actionable, how-to implementation factors for ensuring chronic, preventive, and acute care for patients with diabetes. Employing an innovative Rapid Data Collection and Reporting methodology, teams will rapidly collect, analyze, and share data to accelerate dissemination of customized feedback to FQHC leaders and to inform adaptation and implementation of the iPATH practice transformation.

Aim 2. Implement a multi-level, multi-component, technology-enabled practice transformation strategy to improve type 2 diabetes for patients at 8 multi-clinic FQHCs. Teams will adapt, tailor, implement, test, and spread our practice transformation strategy across FQHCs located in California, Massachusetts, Ohio, and Puerto Rico. The iPATH implementation approach will be modularized and customizable to accommodate organizational readiness, patient needs, and social contexts, tailoring practice transformation efforts to each unique FQHC.

Aim 3. Comprehensively evaluate the iPATH implementation approach with a hybrid type 2 study, including a stepped wedge cluster randomized trial. Including formative, process, and summative evaluation elements guided by the Exploration-Preparation-Implementation-Sustainment model, the study will evaluate impact of practice transformation and identify process elements affecting implementation effectiveness. Analyses will leverage the unique advantage of FQHC data.

ELIGIBILITY:
Inclusion Criteria:

* Two largest clinic sites in multi-clinic FQHCs operating in or near Massachusetts, Ohio, California, Puerto Rico
* We will prioritize FQHCs performing in the lower half of the distribution for A1c control, as these FQHCs have greater room for improvement.

Exclusion Criteria:

* FQHCs that have a patient population comprised of more than 80% children
* FQHCs that have a patient population multiplied by the FQHC's diabetes prevalence in the lowest 10% of all the clinics
* FQHCs that have fewer than 5,000 or more than 50,000 patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119680 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | Before and after 1-year practice transformation period
  Percent poorly controlled diabetes (A1c>9%)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Board of Trustees of the Leland Stanford Junior University, Stanford, California
  - President and Fellows of Harvard College, T.H. Chan School, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
- Impactivo, LLC., San Juan, Puerto Rico, Puerto Rico